CLINICAL TRIAL: NCT04026386
Title: A Center Based Early Intervention Program For Preschoolers With Developmental Disorders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: John & Marcia Goldman Foundation (Unknown)
Responsible Party: Principal Investigator, Antonio Hardan, Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-52348
Record Dates: First submitted 2019-07-17; First posted 2019-07-19 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Development Disorder, Child; Developmental Disability; Development Delay; Autism Spectrum Disorder
MeSH Terms: conditions — Developmental Disabilities; Learning Disabilities; Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Center Based or In-Home Early Intervention Program (Experimental)
  Interventions: Behavioral: Center Based or In Home Early Intervention Program

INTERVENTIONS:
Behavioral: Center Based or In Home Early Intervention Program — This is a 12-week early intervention program that will include 12 weekly hours of treatment in an intensive center-based preschool environment or in home to treat social communication deficits in children with developmental disorders.

SUMMARY:
The purpose of this study is to examine the effectiveness of a 12-week early intervention program that will include 12 weekly hours in an intensive center-based preschool environment or in the home to treat social communication deficits in children with developmental disorders. The study will include children with developmental disorders, such as Autism Spectrum Disorder, neurogenetic disorders, or intellectual disability.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Developmental Disorder, such as Autism Spectrum Disorder, neurogenetic disorder, or intellectual disability, based on clinical interview;
* Boys and girls between 2.0 years and 5.11 years at time of enrollment;
* Ability to participate in the testing procedures to the extent that valid standard scores can be obtained.

Exclusion Criteria:

* Current or lifetime diagnosis of severe psychiatric disorder (e.g., bipolar disorder, etc.);
* Lack of availability during program hours.

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Estimated)
Dates: Start 2019-10-19 (Actual); Primary Completion 2034-12-30 (Estimated); Study Completion 2034-12-30 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Parent Rated Social Responsiveness Scale, 2nd Edition (SRS-2) T-Score After Treatment. | Baseline, 12 Weeks
  Social Responsiveness Scale, 2nd Edition (SRS) scores measure social abilities with lower scores meaning better social abilities. (T-Score Range: 37- above 90 )

SECONDARY OUTCOMES:
Change From Baseline in Parent Rated Repetitive Behavior Scale Revised (RBS-R) Scores During Treatment. | Baseline, 12 Weeks
  Higher scores on the Repetitive Behavior Scale- Revised mean higher levels of repetitive and restricted behaviors. (Raw Score Total Range: 0 - 129)
Change From Baseline in Parent Rated Stanford Social Dimension Scale (SSDS) Scores During Treatment. | Baseline, 12 Weeks
  Higher Scores on the Stanford Social Dimension Scale mean better social functioning and lower scores mean worse social functioning (Range: 58-290).
Change From Baseline in Parent Rated Vineland Adaptive Behavior Scale- 3 (VABS-3) Scores During Treatment. | Baseline, 12 Weeks
Change From Baseline in Parent Rated Short Sensory Profile Questionnaire (SSPQ) Scores During Treatment. | Baseline, 12 Weeks
Change From Baseline in Parent Rated General Self Efficacy Scale (GSES) Scores During Treatment. | Baseline, 12 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Hardan, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No